CLINICAL TRIAL: NCT00344591
Title: Ecosystems Therapy for Men Reintegrating Into Their Family
Brief Title: Effectiveness of Structured Ecosystems Therapy for Reducing HIV Risk Behaviors and Improving Treatment Adherence in HIV Infected Men Released From Prison
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: R01MH067495 (NIH); R01MH067495 (NIH); DAHBR 9A-ASI
Record Dates: First submitted 2006-06-23; First posted 2006-06-27 (Estimated); Last update posted 2015-07-24 (Estimated); Status verified 2015-07

CONDITIONS: HIV Infections; Acquired Immunodeficiency Syndrome
Keywords: HIV; AIDS
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome

ARMS (2):
- Tailored SET program (Experimental): tailored SET program for reducing sexual and drug-related HIV transmission risk factors and increasing HIV treatment adherence in HIV infected men who have recently been released from prison
  Interventions: Behavioral: Structured Ecosystems Therapy (SET)
- Individually focused therapy (Active Comparator): Individually focused therapy program for reducing sexual and drug-related HIV transmission risk factors and increasing HIV treatment adherence in HIV infected men who have recently been released from prison
  Interventions: Behavioral: Individually tailored intervention

INTERVENTIONS:
Behavioral: Structured Ecosystems Therapy (SET)
  Arms: Tailored SET program
Behavioral: Individually tailored intervention
  Arms: Individually focused therapy

SUMMARY:
This study will evaluate the effectiveness of Structured Ecosystems Therapy (SET), a form of therapy that includes family and caregivers, at reducing HIV transmission risk behaviors and improving treatment adherence in HIV infected men newly released from prison.

DETAILED DESCRIPTION:
Individuals in prison are four times more likely to have HIV or AIDS as compared to non-incarcerated people. Once HIV infected individuals are released from prison, they have a high risk of transmitting HIV to their sexual or needle-sharing partners. Therefore, it is important to encourage HIV risk reduction behavior among such inmates who are nearing release from prison. SET is a therapy program that mobilizes family and caregivers as a way to support and encourage behavior change within an individual. This study will use a tailored SET program to meet the specific needs of prisoners who are infected with HIV. The purpose of the study is to compare the effectiveness of the tailored SET program versus an individually focused therapy program at reducing sexual and drug-related HIV transmission risk factors and increasing HIV treatment adherence in HIV infected men who have recently been released from prison.

This 12-month study will enroll HIV infected men who are being released from the California Medical Facility Prison in Vacaville, California or the San Quentin State Prison in Marin County, California. Participants will meet with study recruiters while in prison and complete questionnaires to assess sexual and drug-related HIV transmission risk behaviors and treatment adherence; they will also participate in a health education session. Participants will then be randomly assigned to either a 4-month tailored SET program or a 4-month individually focused therapy program. All participants will meet with study counselors twice while still in prison, and then weekly during the first 4 months following release from prison. Participants in the SET program will work with study counselors to tailor the program to meet their individual needs. Therapy sessions will be designed to restructure interactions and communication patterns between the participant and his support network; main goals will include reducing sexual and drug-related risk behaviors and improving HIV treatment adherence. Participants in the individually focused therapy program will focus on harm reduction, goal setting, and motivational enhancement. HIV transmission risk behaviors and treatment adherence will be assessed with surveys administered at Months 4, 8, and 12 for all participants.

ELIGIBILITY:
Inclusion Criteria:

* HIV infected
* Scheduled to be released from the California Medical Facility Prison in Vacaville, California or from San Quentin State Prison in Marin County, California between 21 to 90 days following study entry
* Speaks English or Spanish
* Able to provide contact information for at least one adult who will be living in the area and is able to participate in the study

Exclusion Criteria:

* Participation in the pilot study or previous enrollment in the study
* Release into another correctional facility or other restricted environment (after the initial release from prison) that would prevent participation in the study for more than 2 weeks (e.g., drug treatment program that does not allow visitors)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2005-01; Primary Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
HIV transmission risk behaviors | 12 months
HIV-related medical adherence | 12 months

SECONDARY OUTCOMES:
Mediators of HIV transmission risk reduction and medical adherence | 12 months
Recidivism to prison | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Olga Grinstead, PhD, MPH, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States